CLINICAL TRIAL: NCT03918772
Title: Clinical Determinants in Perioperative Allergic Immediate Hypersensitivity
Brief Title: Clinical Determinants and Perioperative Allergic Reactions (CADECAP Study)
Acronym: CADECAP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-043
Record Dates: First submitted 2019-03-12; First posted 2019-04-18 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-03

CONDITIONS: Hypersensitivity, Immediate; Perioperative Period
Keywords: Anaphylaxis; Epinephrine; Hypersensitivity, Immediate; Morbidity; Mortality; Perioperative Period; Skin Tests; Tryptases
MeSH Terms: conditions — Hypersensitivity, Immediate; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perioperative immediate hypersensitivity: Patients having experienced perioperative immediate hypersensitivity

SUMMARY:
The clinical presentation of perioperative allergic and non-allergic clinical reactions is often considered undistinguishable while the accurate analysis of clinical cases shows striking clinical differences which might be predictive of the etiological diagnosis (allergic versus non-allergic).

The four-step Ring and Messmer clinical scale helps to guide acute management of immediate hypersensitivity accordingly to the clinical presentation although this scale does not take into account the mechanism involved (i.e. allergic versus non-allergic). Non-allergic clinical reactions are usually non-life-threatening and may, sometimes, spontaneously resolve in contrast to allergic reactions which are mainly severe and life-threatening conditions, typically called anaphylaxis.

The cornerstones of anaphylaxis management are fluid therapy and epinephrine. However, poor outcome has been reported as a result of delayed treatment and/or inappropriate management of perioperative anaphylaxis.

DETAILED DESCRIPTION:
The main objectives of this study are to: i) characterize the clinical and paraclinical determinants of IgE-mediated allergy that could be correlated to the ultimate diagnosis; and ii) elaborate a decision-making algorithm for clinical patterns identification of perioperative allergic reactions to guide acute management, thus potentially decreasing the related morbidity and mortality.

The secondary objectives are to: i) suggest a modification of the Ring and Messmer scale according to the phenotypes involved; ii) identify the clinical characteristics of isolated non-allergic bronchospasm; iii) compare the most frequent agents involved in perioperative IgE-mediated allergy to those reported in the international studies; iv) identify the negative predictive values of skin tests in allergic and non-allergic patients; v) compare the therapeutic modalities used to those recommended in the literature; vi) describe the cases of morbidity and mortality and identify the potential risk factors.

The Ring and Messmer scale is used to quote the clinical features occurring in drug- or latex-induced immediate hypersensitivity and has been adapted to the perioperative setting as follows:

Grade I: Muco-cutaneous signs only (generalized erythema and/or extensive urticaria and/or angioedema) Grade II: Mucocutaneous signs, hypotension, tachycardia and/or moderate bronchospasm Grade III: Mucocutaneous signs, cardiovascular collapse, tachycardia or bradycardia, bronchospasm, digestive signs Grade IV: Cardiac arrest Grade V: Death

Perioperative immediate hypersensitivity reaction requires further allergologic assessment.

The allergologic assessment is performed a few weeks after the reaction to confirm or disprove an allergic mechanism behind the reaction (i.e. allergy versus non-allergy), and to identify culprit agent(s) and safe drugs, including suitable alternatives. It is based on the review of the details of the reaction along with histamine and/or tryptase levels and specific Immunoglobulin E levels (when available) and skin tests results.

Plasma histamine and/or tryptase levels and Immunoglobulin E levels are measured at the time of the reaction. Acute tryptase levels are compared to baseline tryptase measured at least 24 hours after the reaction or when the patient is referred for allergological investigation. Skin tests, including prick-tests and intradermal tests, are performed during the allergological assessment.

ELIGIBILITY:
Inclusion criteria:

* Patients having experienced a perioperative immediate hypersensitivity (including the obstetrical setting) according to one grade of the Ring and Messmer clinical scale, for whom:
* The clinical history is known and has been related to perioperative immediate hypersensitivity;
* The biological assessment including plasma histamine and/or tryptase (and serum IgE when available) was performed after the onset of immediate hypersensitivity according to current guidelines;
* The allergological assessment including skin tests performed by the collaborators of this study was carried out according to current guidelines in surviving patients

Exclusion criteria:

• Patients who decline to be involved in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having experienced a perioperative immediate hypersensitivity where the allergological assessment was performed by the collaborators of this study
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Identification of the predictive muco-cutaneous signs of perioperative allergic immediate hypersensitivity as assessed by the Ring and Messmer clinical scale | From date of the perioperative clinical reaction up to 6 hours
  muco-cutaneous signs (generalized erythema and/or extensive urticaria and/or angioedema)
Identification of the predictive heart rate of perioperative allergic immediate hypersensitivity as assessed by the Ring and Messmer clinical scale | From date of the perioperative clinical reaction up to 6 hours
  heart rate (beat/min.)
Identification of the predictive arterial pressure of perioperative allergic immediate hypersensitivity as assessed by the Ring and Messmer clinical scale | From date of the perioperative clinical reaction up to 6 hours
  arterial pressure (mmHg)
Identification of the predictive upper gastrointestinal symptoms of perioperative allergic immediate hypersensitivity as assessed by the Ring and Messmer clinical scale | From date of the perioperative clinical reaction up to 6 hours
  digestive signs (vomiting)
Identification of the predictive lower gastrointestinal symptoms of perioperative allergic immediate hypersensitivity as assessed by the Ring and Messmer clinical scale | From date of the perioperative clinical reaction up to 6 hours
  digestive signs (diarrhea)
Identification of recurrence of perioperative allergic immediate hypersensitivity as assessed by the Ring and Messmer clinical scale | From date of the perioperative clinical reaction up to 6 hours
  recurrence of symptoms following a symptom-free response

SECONDARY OUTCOMES:
Drugs involved in adverse reactions as assessed by the Ring and Messmer clinical scale | From date of the perioperative clinical reaction and up to 100 months
  To identify the drugs involved in the onset of perioperative allergic clinical reactions and compare our results to those provided in the different international epidemiologic studies regarding perioperative immediate hypersensitivity.
Negative predictive values of skin tests in allergic and non-allergic patients | Up to 5 years after the allergologic follow-up
  Negative skin-tested agents administered according to the results of allergological follow-up during subsequent anesthetics in allergic and non-allergic patients
Participants with treatment-related adverse events as assessed by by CTCAE v4.0 and fluid therapy | Through study completion, an average of 2 years
  To identify the number of patients who received fluid therapy (volume, type) in allergic hypersensitivity
participants with treatment-related adverse events as assessed by CTCAE v4.0 and vasoconstrictive agents | Through study completion, an average of 2 years
  To identify the number of patients who received vasoconstrictive agents (ephedrine, neosynephrine, epinephrine, norepinephrine) and corresponding cumulative doses
participants with treatment-related adverse events as assessed by CTCAE v4.0 and salbutamol and/or steroids | Through study completion, an average of 2 years
  To identify the number of patients who received salbutamol, steroids and corresponding doses
Participants with treatment-related adverse events as assessed by CTCAE v4.0 and intensive care unit admission | Through study completion, an average of 2 years
  To identify the number of patients who were admitted in intensive care unit
Participants with treatment-related adverse events as assessed by CTCAE v4.0 and morbidity | Through study completion, an average of 2 years
  To report the morbidity cases including cardiac and/or renal and/or hepatic and/or neurologic failure(s) after perioperative allergic immediate hypersensitivity
Participants with treatment-related adverse events as assessed by CTCAE v4.0 and mortality | Through study completion, an average of 2 years
  To report the mortality cases after perioperative allergic immediate hypersensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Dewachter, M.D., Ph.D., Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique-Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No